CLINICAL TRIAL: NCT01434225
Title: NEMO1: An Open Label Exploratory Dose Finding and Pharmacokinetic Clinical Trial of Bumetanide for the Treatment of Neonatal Seizure Using Medication Off-patent
Brief Title: NEMO1:NEonatal Seizure Using Medication Off-patent
Acronym: NEMO1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Only For Children Pharmaceuticals (Industry); Cork University Hospital (Other); UMC Utrecht (Other); Helsinki University Central Hospital (Other); Hôpital Necker-Enfants Malades (Other); The Leeds Teaching Hospitals NHS Trust (Other); Karolinska University Hospital (Other); University College London Hospitals (Other); Uppsala University Hospital (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08NR26
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Neonatal Seizures
Keywords: Neonatal seizures; Hypoxic Ischemic Encephalopathy; Electroencephalography; Bumetanide
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Bumetanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bumetanide (Experimental): Bumetanide - Standard Phenobarbital plus either 0.05 mg/kg,0.1 mg/kg, 0.2 mg/kg, or 0.3 mg/kg of bumetanide as determined by the the dose escalation design Maximum dose allowed is 0.3mg/kg given up to 4 times at 12 hourly intervals (total of 1.2mg/kg).
  Interventions: Drug: Bumetanide

INTERVENTIONS:
Drug: Bumetanide — Bumetanide - Standard Phenobarbital plus either 0.05 mg/kg,0.1 mg/kg, 0.2 mg/kg, or 0.3 mg/kg of bumetanide as determined by the the dose escalation design Maximum dose allowed is 0.3mg/kg given up to 4 times at 12 hourly intervals (total of 1.2mg/kg).

SUMMARY:
NEMO is a multicentre pan European clinical trial with the aim to develop new treatment strategies for the treatment of neonatal seizures using the loop diuretic bumetanide. There is evidence that bumetanide improves GABAergic function of the current standard drug, phenobarbitone. Bumetanide has been used as a diuretic in term and preterm babies for around thirty years. This trial should confirm that Bumetanide in addition to standard treatment will result in better seizures control.

ELIGIBILITY:
Inclusion Criteria:-

* Male or female term baby with gestational age of 37-43 weeks and postnatal age <48 hours
* One or more of the following:
* APGAR score < 5 at 5 mins.
* Umbilical cord or first arterial blood sample pH < 7.1 or base deficit >16 mmol/L.
* Postnatal resuscitation still required 10 minutes after birth

  * Clinically evolving encephalopathy
  * Received one dose of standard anticonvulsive therapy (phenobarbitone,20mg/kg) for clinical or electrographic seizures.
  * EEG: equal to or more than 3 min cumulative seizures, or 2 or more seizures of >30 sec duration over 2 hr period within first 48 hr of life
  * Written informed consent of parent or guardian.
  * EEG monitoring has commenced within the first 48 hours of birth.

Exclusion Criteria:

* Suspected or confirmed brain malformation, inborn error of metabolism,genetic syndrome, or major congenial malformation
* Congenital (in utero) infection (TORCH).

  * Babies who have received diuretics such as furosemide or bumetanide in routine clinical management within the last 24 hours.
  * Total serum bilirubin > 15 mg/dl (255 micromol/l) at inclusion.
  * On any other anticonvulsive medication other than phenobarbitone or bolus of midazolam / pentobarbitone for intubation.
  * Anuria/renal failure defined as serum creatinine > 200 micromol/l.
  * Severe electrolyte depletion (Na <120 mmol/L, K <3.0 mmol/L)

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Optimal dose finding | 6 months
  The optimal dose is defined as achieving effective seizure reduction:
  * Reduction of electrographic seizure (measuresd by EEG) burden by >80% during the 3rd and 4th hour after the first bumetanide administration compared to a 2 hour epoch prior to Bumetanide administration.
  * No need for rescue AED within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Pressler, Dr, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (7):
- Cork University Maternity Hospital, Cork, Ireland
- Netherlands (2):
  - Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam
  - University Medical Centre Utrecht, Utrecht
- Sweden (2):
  - Karolinska Institutet and University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - Leeds General Infirmary, Leeds
  - University College London Hospitals NHS Foundation Trust, London

REFERENCES:
- [Derived] Pressler RM, Boylan GB, Marlow N, Blennow M, Chiron C, Cross JH, de Vries LS, Hallberg B, Hellstrom-Westas L, Jullien V, Livingstone V, Mangum B, Murphy B, Murray D, Pons G, Rennie J, Swarte R, Toet MC, Vanhatalo S, Zohar S; NEonatal seizure treatment with Medication Off-patent (NEMO) consortium. Bumetanide for the treatment of seizures in newborn babies with hypoxic ischaemic encephalopathy (NEMO): an open-label, dose finding, and feasibility phase 1/2 trial. Lancet Neurol. 2015 May;14(5):469-77. doi: 10.1016/S1474-4422(14)70303-5. Epub 2015 Mar 10. PMID 25765333